CLINICAL TRIAL: NCT01997502
Title: Prospective Observational Study Characterizing Noninvasive Hemoglobin (SpHb) Measured With Pulse CO-Oximetry Technology in a Variety of Surgical Cases
Brief Title: Accuracy of Pulse CO-Oximetry Technology in Characterizing Noninvasive SpHb
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 494171
Record Dates: First submitted 2013-11-01; First posted 2013-11-28 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2024-11

CONDITIONS: Surgery; Hemoglobin
Keywords: Hemoglobin; Non-invasive
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Pulse CO-Oximetry Technology — In addition to the standard pulse oximeter used for clinical care, up to six SpHb finger sensors will be applied to the patient. Additional sensors may also be applied to the forehead, neck, chest and ears.
  Masimo FDA cleared pulse CO-Oximeter devices: Radical-7, Rad-87, Rad-57, Pronto, Pronto-7, for the noninvasive measurement of SpO2, PR, PI, PVI, SpCO, SpMet, and SpHb, total hemoglobin and respiratory rate.
  No treatment decisions will be made based on the new technology and no extra medical procedures are required for the study.
Other: Blood draw — 4mL arterial blood samples (up to 1 per hour), outside standard of care, are drawn throughout the surgical procedure and sent to UCDMC lab/Masimo lab for analysis.

SUMMARY:
This protocol is a request from Masimo to assist in the collection of data to be used to further refine the accuracy of the monitor's algorithm.

DETAILED DESCRIPTION:
The specific aim of this study is to collect data to characterize Masimo's noninvasive Rainbow SpHb technology during surgeries. The purpose is to compare Masimo Rainbow technology to arterial blood samples taken during surgery. Hemoglobin concentrations in the arterial blood samples will be measured using standard blood analyzers on site and/or the sponsor's laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery requiring intra-arterial pressure monitoring

Exclusion Criteria:

* Age less than 18 years
* Pregnancy
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 621 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Comparison of Masimo Rainbow technology to arterial blood samples taken during surgery | Five year
  Correlation between standard, lab-based, hemoglobin measurement and concurrent SpHb.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Fleming, M.D., Ph.D., Principal Investigator — Professor, Director, Cardiovascular and Thoracic Anesthesiology
Locations (1):
- UC Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-the-accuracy-of-experimental-pulse-co-oximetry-technology-for-noninvasive-hemoglobin-sphb-measurements-766867/